CLINICAL TRIAL: NCT04346589
Title: A Pilot Study to Explore the Efficacy and Safety of Rescue Theraphy With Antibodies From Convalescent Patients Obtained With Double -Filtration Plasmapheresis (DFPP) and Infused in Critically Ill Ventilated Patients With Coronavirus Disease 2019 (COVID-19)
Brief Title: Convalescent Antibodies Infusion in Critically Ill COVID 19 Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed prematurely because the hyperimmune plasma have expired
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Aferetica - Italy (BO) (Unknown)
Responsible Party: Principal Investigator, Piero Luigi Ruggenenti, Director, Unit of Nephrology, A.O. Ospedale Papa Giovanni XXIII
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFPP COVID 19
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Pneumonia, Ventilator-Associated; Coronavirus Infection
Keywords: Pneumonia COVID 19 ventilator-dependent; COVID19; Double-filtration plasmapheresis; Convalescent antibodies
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antibodies (immunoglobulins) infusion (Experimental): Anti-coronavirus antibodies obtained with double-filtration plasmapheresis (DFPP )from convalescent patients.
  Interventions: Biological: Anti-coronavirus antibodies (immunoglobulins)obtained with DFPP from convalescent patients

INTERVENTIONS:
Biological: Anti-coronavirus antibodies (immunoglobulins)obtained with DFPP from convalescent patients — Antibodies obtained from consenting convalescent donors will be administered to ten consecutive patients who fulfill the inclusion criteria . Convalescent antibodies will be obtained with one DFPP procedure from consenting donors and infused in one critically ill, ventilated patient with COVID 19 pneumonia.

SUMMARY:
The 2019 outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 or COVID 19), which originated in Wuhan, China, has become a major concern all over the world.

Convalescent plasma or immunoglobulins have been used as a last resort to improve the survival rate of patients with SARS whose condition continued to deteriorate despite any attempted treatment.. Moreover, several studies showed a shorter hospital stay and lower mortality in patients treated with convalescent plasma than those who were not treated with convalescent plasma. Evidence shows that convalescent plasma from patients who have recovered from viral infections can be used effectively as a treatment of patients with active disease.

The use of solutions enriched of antiviral antibodies has several important advantages over the convalescent plasma including the high level of neutralizing antibodies supplied. Plasma-exchange is expensive and requires large volumes of substitution fluid. Albumin is better tolerated and less expensive, but exchanges using albumin solutions increase the risk of bleeding because of progressive coagulation factor depletion. With either albumin or fresh frozen plasma, increasing the risk of cardiovascular instability in the plasma donor and in the recipient, which can be detrimental in a critically ill patient with COVID 19 pneumonia.

The aforementioned limitations of plasma therapy can be overcome by using selective apheresis methods, such as double-filtration plasmapheresis (DFPP).DFPP is a modality of plasma purification that performs an initial plasma separation from blood, and the subsequent separation of specific molecules, on the basis of their specific molecular weight (cut-off), by using a fractionation filter. The Fractionation Filter 2A20, because of its membrane sieving cut-off, retains larger molecules and returns plasma along with smaller molecules to the circulation, including the major part of the albumin. The selection of the membrane 2A20 is related to the appropriate Sieving Coefficient for IgG that allows to efficiently collect antibodies from patients which are recovered from COVID-19, with negligible fluid losses and limited removal of albumin. The total amount of antibodies obtained during one DFPP session exceeds by three to four times the total amount provided to recipients with one unit of plasma obtained during one plasma-exchange session from one COVID-19 convalescent donor. This should result in more effective viral inhibition and larger benefit for the patient achieved with one unit of enriched immunoglobulin solution obtained with DFPP than with one unit of plasma obtained with plasma exchange.

These observations provide the background for a pilot study aimed to explore whether the infusion of antibodies obtained with one single DFPP procedure from voluntary convalescent donors could offer an effective and safe therapeutic option for critically ill patients with severe coronavirus (COVID-19) pneumonia requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

Plasma Ig Donors

* Adult (>18 and <65-yr-old) men and women
* Convalescent donor who recovered from COVID 19 from at least 14 days according to the clinical and laboratory criteria defined by the Consiglio Superiore di Sanità on February 20, 2019 ("The recovered patient is the one who resolves the symptoms of COVID-19 infection and who is negative in two consecutive tests for the search for SARS-Cov-2, performed 24 hours apart") with the exceptions mentioned in the attached derogation (that is "no upper age limit to donation provided there are no clinical contraindications to the procedure and independent of documented evidence of two negative tests for SARS-Cov 2 naso-faringeal contamination")
* Male or female donor; if female only if nulliparous; in both cases with a negative history of blood component transfusions
* Careful clinical evaluation of the patient-donor with particular reference to the criteria established by current legislation to protect the health of the donor who donates by apheresis
* Presence of adequate levels of neutralizing anti-SARS-COV-2 antibodies;
* Biological qualification test negative defined by current indications (performed at SIMT of HPG23)
* Test negative for: HAV RNA, HEV RNA, PVB19 DNA (performed at HPG23)
* Informed consent

Recipients

* Adult (>18-yr-old) men and women
* COVID-19 pneumonia diagnosed by standard criteria
* Need of ventilator support
* Informed consent for participation in the study (critically ill patients will be unable to provide consent. Consent will be oral if a written consent will be impossible. If the subject is incapable of giving an informed consent and an authorized representative is not available without a delay that would, in the opinion of the Investigator, compromise the potential life-saving effect of the treatment this can be administered without consent. Consent to remain in the research should be sought as soon as the conditions of the patient will allow it).
* <48 hours of mechanical ventilation

Exclusion Criteria:

* >48 hour mechanical ventilation
* Patient being treated with other anti-COVID-19 experimental treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Number of mechanical ventilation days. | Through study completion, an average of 6 months.

SECONDARY OUTCOMES:
Survival | Through study completion, an average of 6 months.
Shift to Continuous Positive Airway Pressure (CPAP) ventilation | Through study completion, an average of 6 months.
Referral to a sub-intensive care unit or discharge | Through study completion, an average of 6 months.
Viral titer | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
Anti COVID 19 IgG antibodies | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
Anti COVID 19 IgM antibodies | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
C5a concentration | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
  Marker of complement activation in plasma.
C3a concentration | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
  Marker of complement activation in plasma.
Serum C5b-9 concentration | Changes from before Ig administration, one day and one week after Ig administration and every week after discharge from the intensive care unit through study completion, an average of 6 months.
  Marker of complement activation in plasma.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - IRFMN - Clinical Research Center for Rare Diseases, Ranica, BG
  - ASST HPG23 - Unit of Nephrology, Bergamo
  - ASST Papa Giovanni XXIII - Microbiology and Virology Unit, Bergamo
  - Asst Pg23 - S.I.M.T, Bergamo
  - ASST-PG23 - Intensive Care Unit, Bergamo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Curto D, Tomatis F, Gastoldi S, Galbusera M, Noris M, Raimondi F, Lorini FL, Falanga A, Marchetti M, Remuzzi G, Ruggenenti P. Case Report: Effects of Anti-SARS-CoV-2 Convalescent Antibodies Obtained With Double Filtration Plasmapheresis. Front Immunol. 2021 Jun 30;12:711915. doi: 10.3389/fimmu.2021.711915. eCollection 2021. PMID 34276706